CLINICAL TRIAL: NCT03106909
Title: Feasibility and Reliability of Pulmonary Computed Tomography as a Radiological Reference Standard for Evaluating Chest X-ray and Candidate Biomarkers in Suspected Pneumonia Complicating Stroke
Brief Title: Pulmonary CT in Pneumonia Complicating Stroke
Status: Completed | Type: Observational
Sponsor: Natalie Garratt (Other)
Responsible Party: Sponsor-Investigator, Natalie Garratt, Research & Development Lead, Northern Care Alliance NHS Foundation Trust
Organization: Northern Care Alliance NHS Foundation Trust (Other)
Other Study IDs: 213436
Record Dates: First submitted 2017-02-01; First posted 2017-04-11 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Pneumonia
Keywords: stroke; pneumonia; biomarkers; pulmonary CT
MeSH Terms: conditions — Stroke; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: pulmonary computed tomography (CT) — Pulmonary CT imaging

SUMMARY:
Pneumonia commonly complicates stroke and has a profound impact on clinical outcomes. Accurate and timely diagnosis of pneumonia complicating stroke remains a major challenge as several issues potentially confound diagnosis. Chest X-ray (CXR), a central component in the diagnostic work-up, may have limited utility in the early stages as they are often of suboptimal quality, and infrequently confirm typical diagnostic infiltrates. Blood biomarkers of the stress-immune response have received considerable attention, but interpretation has been limited by differing methodologies, including definition of pneumonia. Bacterial organisms in the oral cavity may also be of relevance as biomarkers of post-stroke pneumonia. Major challenges facing frontline clinicians are therefore whether to initiate antibiotics; if so, when and for how long. These issues have antibiotic stewardship implications for clinicians in terms of potential for under-treatment or over-treatment with antibiotics based on CXR appearances.

Pulmonary Computed Tomography (CT) could be of value as a radiological reference standard when pneumonia is suspected after stroke, and enable more rigorous evaluation of the diagnostic performance of CXR (and other candidate biomarkers) to inform decision-making when pneumonia is suspected.

The overall primary aim is therefore to investigate the feasibility and reliability of using pulmonary CT as a radiological reference standard for evaluating suspected pneumonia complicating stroke. The secondary aims are to explore the diagnostic accuracy of CXR and blood biomarkers (index tests) when pneumonia is suspected during hospital admission after stroke using pulmonary CT as a reference standard.

DETAILED DESCRIPTION:
Pneumonia is a frequent complication of stroke, particularly within the first few days. The risk of pneumonia is increased in patients who are older, have a more severe stroke and in those who have swallowing problems as a result of their stroke. Patients who develop pneumonia have a higher risk of death and longer hospital stay. The diagnosis of pneumonia is not always easy, but it is important to identify pneumonia early in order to begin the most appropriate treatment in a timely fashion and avoid giving antibiotics unnecessarily. Chest x-ray, the standard test undertaken when pneumonia is suspected, infrequently shows changes and is of limited value.

Pulmonary Computed Tomography (CT) scans can be used to image the lungs in more detail than a standard chest xray. The Investigators plan to assess if it is feasible to perform pulmonary CT imaging in stroke patients within 48 hours of symptoms and who may be acutely unwell. The Investigators will also investigate how reliable CT is at diagnosing pneumonia by asking different x-ray doctors to review the scans. Comparing the result of the pulmonary CT imaging to the chest x-ray will allow assessment of their utility for the diagnosis of pneumonia. The Investigators will also record whether the CT informs clinical management e.g. stopping antibiotics if pneumonia is excluded.

Blood samples will be collected for measurement of inflammatory markers and mouth swabs will measure types of bacteria. The analysis will be conducted at Salford Royal NHS Foundation Trust (SRFT) and using new cutting-edge techniques performed by collaborators at ThermoFisher and Manchester Collaborative Centre for Inflammation Research. The Investigators will assess how useful these inflammatory proteins are in pneumonia diagnosis compared to the pulmonary CT scans. This research will help the Investigating team design larger studies to diagnose pneumonia earlier and more accurately, enabling more effective use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient in SRFT or RSUH with diagnosis of stroke current admission
* Within 24h of clinically suspected pneumonia occurring after admission
* Aged ≥18y
* Provision of informed consent from participant or personal consultee
* Able to undergo pulmonary CT within next 48h

Exclusion Criteria:

* Treatment for lower respiratory tract infection (LRTI) completed within the preceding month
* Mechanical ventilation planned or anticipated imminently
* End-of-life care planned or anticipated imminently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient stroke service at Salford Royal Foundation Trust (SRFT) and Royal Stoke University Hospital (RSUH)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Proportions of eligible participants from screening; eligible participants declining participation (and reasons) | 18 months
Proportion of participants undergoing pulmonary CT | 18 months
  Participants scanned and reasons for not scanning

SECONDARY OUTCOMES:
Proportion of consenting participants undergoing repeat CXR when indicated | 18 months
Proportion with changes consistent with pneumonia on CXR; proportion with changes consistent with pneumonia on pulmonary CT | 18 months
Proportion participants with changes consistent with pneumonia on pulmonary CT | 18 months
Characteristics and distribution of radiological changes consistent with pneumonia on pulmonary CT | 18 months
  Using standard assessments of diagnostic accuracy, including sensitivity, specificity, positive and negative predictive values
Spectrum of additional radiological findings on pulmonary CT | 18 months
Inter-rater reliability of CXR; and pulmonary CT interpretation | 3 months
  Inter-rater reliability of the CXR reports will be evaluated using k statistics and the Bland and Altman method
Inter-rater reliability of pulmonary CT interpretation | 3 months
  Inter-rater reliability of the pulmonary CT reports will be evaluated using k statistics and the Bland and Altman method
Proportion of participants with confirmed pneumonia | 18 months
  Confirmed pneumonia is defined as meeting the PISCES clinical criteria AND with changes of pneumonia on pulmonary CT, agreed by an adjudication panel
Estimate and confidence intervals of sensitivity and specificity of CXR | 3 months
  Using diagnostic odds ratio for CXR singly and with repeat CXR where indicated clinically
Estimate and confidence intervals of sensitivity and specificity of C-reactive protein (CRP) markers | 18 months
  Using standard assessments of diagnostic accuracy, including sensitivity, specificity, positive and negative predictive values
Estimate and confidence intervals of sensitivity and specificity of procalcitonin (PCT) | 18 months
  Using standard assessments of diagnostic accuracy, including sensitivity, specificity, positive and negative predictive values
Estimate and confidence intervals of sensitivity and specificity of copeptin | 18 months
  Using standard assessments of diagnostic accuracy, including sensitivity, specificity, positive and negative predictive values
Estimate and confidence intervals of sensitivity and specificity of pro-adrenomedullin (Pro-ADM) | 18 months
  Using standard assessments of diagnostic accuracy, including sensitivity, specificity, positive and negative predictive values
Estimate and confidence intervals of sensitivity and specificity of monocyte/ B-cell markers | 18 months
  Using standard assessments of diagnostic accuracy, including sensitivity, specificity, positive and negative predictive values
Characteristics of oral bacterial species | 18 months
  Oral bacterial species will be compared in patients with and without confirmed pneumonia in univariate hypothesis generating analyses
Distribution of oral bacterial species | 18 months
  Oral bacterial species will be compared in patients with and without confirmed pneumonia in univariate hypothesis generating analyses
Number of days of antibiotic treatment | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: CRAIG SMITH, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Salford Royal Nhs Foundation Trust, Salford, Greater Manchester
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers